CLINICAL TRIAL: NCT02090842
Title: Investigating the Acute and Chronic Effects of Dietary Proteins on Markers of Vascular Function, Ambulatory Blood Pressure, Insulin Resistance and Lipid Metabolism.
Brief Title: Milk Proteins, Ambulatory Blood Pressure and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Volac Int. Ltd. (Unknown)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 12/40
Record Dates: First submitted 2013-06-17; First posted 2014-03-18 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension
Keywords: Milk proteins; Blood pressure; Vascular function
MeSH Terms: conditions — Hypertension | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Whey protein isolate (Experimental): Subjects are asked to supplement their habitual diet with 56 g of whey protein isolate a day for 8 weeks.
  Interventions: Dietary Supplement: Whey protein isolate
- Ca-caseinate (Experimental): Subjects are asked to supplement their habitual diet with 56 g of Ca-caseinate a day for 8 weeks.
  Interventions: Dietary Supplement: Ca-caseinate
- Maltodextrin (Other): Subjects are asked to supplement their habitual diet with 54 g of maltodextrin a day for 8 weeks.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Ca-caseinate
  Arms: Ca-caseinate
Dietary Supplement: Maltodextrin
  Arms: Maltodextrin
Dietary Supplement: Whey protein isolate
  Arms: Whey protein isolate

SUMMARY:
Epidemiological studies demonstrated an inverse associations between cardiovascular events and milk and dairy product consumption. Evidence from human intervention studies suggests that both whey and casein may be effective in blood pressure-lowering, however there is limited data on the impact of milk proteins on vascular function. This research aims to compare the potential acute and chronic impacts of the two main milk proteins (whey and casein) with maltodextrin on blood pressure and vascular function. Furthermore, the effects of these proteins on the markers of insulin resistance, lipid metabolism and inflammatory status will also be investigated in 'at-risk' individuals.

This research includes both an acute and chronic intervention study which have been independently powered on the appropriate outcome measures. This has generated different sample size requirements for the two studies (Actual participants on the acute study: n=27, and on the chronic study: n=38).

ELIGIBILITY:
Inclusion Criteria:

* A signed consent form
* Blood pressure: 120/80-159/99
* Age: 30-77 years
* BMI 20-40 kg/m2
* Glucose <7 mmol/l (Not diagnosed with diabetes)
* Chol <8 mmol/l
* TAG <4 mmol/l
* Normal liver and kidney function
* Haemoglobin (>110 g/dl women; 140g/dl men)

Exclusion Criteria:

* Milk allergy, lactose allergy
* Coeliac disease
* Renal, gastrointestinal, respiratory, endocrine, liver disease or cancer
* Surgery in the previous 6 months
* Secondary hypertension
* Excess alcohol consumption (drinking >28 unit/wk man; >21 unit/wk women)
* Smoker
* Vegan
* Taking nutritional supplementation (e.g. fish oil, proteins)
* Anaemia

Ages: 30 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in 24-h ambulatory blood pressure | Chronic study: Baseline and week 8 assessments for the three dietary intervention arms, Acute study: automated ambulatory blood monitor measures every 15 minutes for 3 hours after both meals, then every 30 minutes for day

SECONDARY OUTCOMES:
Changes in vascular reactivity measured by flow-mediated dilation (FMD) | Chronic study: Baseline and week 8 assessments for the two dietary intervention arms, Acute study: determined at 0 (fasted), 180, 300, 420 min
Changes in plasma lipids | Chronic study: Baseline and week 8 assessments for the two dietary intervention arms, Acute study: fasted and postprandial
Changes in markers of insulin resistance | Chronic study: Baseline and week 8 assessments for the two dietary intervention arms, Acute study: fasted and postprandial
Changes in inflammatory markers | Chronic study: Baseline and week 8 assessments for the two dietary intervention arms, Acute study: fasted and postprandial
Changes in arterial stiffness measured by pulse wave analysis (PWA) | Chronic study: Baseline and week 8 assessments for the two dietary intervention arms, Acute study: determined at 0 (fasted), 180, 300, 420 min
Changes in arterial stiffness measured by digital volume pulse (DVP) | Chronic study: Baseline and week 8 assessments for the two dietary intervention arms, Acute study: determined at 0 (fasted), 180, 300, 420 min

OTHER OUTCOMES:
Handgrip strength measurement | Chronic study: Baseline and week 8 assessments for the two dietary intervention arms
Metabonomics | Chronic study: Baseline and week 8 assessments for the two dietary intervention arms; Acute study: fasted and postprandial

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Lovegrove, BSc, PhD, RNutr, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, Berks, United Kingdom

REFERENCES:
- [Background] Pal S, Ellis V. Acute effects of whey protein isolate on blood pressure, vascular function and inflammatory markers in overweight postmenopausal women. Br J Nutr. 2011 May;105(10):1512-9. doi: 10.1017/S0007114510005313. Epub 2011 Jan 28. PMID 21272399
- [Background] Pal S, Ellis V. The chronic effects of whey proteins on blood pressure, vascular function, and inflammatory markers in overweight individuals. Obesity (Silver Spring). 2010 Jul;18(7):1354-9. doi: 10.1038/oby.2009.397. Epub 2009 Nov 5. PMID 19893505
- [Derived] Fekete AA, Giromini C, Chatzidiakou Y, Givens DI, Lovegrove JA. Whey protein lowers blood pressure and improves endothelial function and lipid biomarkers in adults with prehypertension and mild hypertension: results from the chronic Whey2Go randomized controlled trial. Am J Clin Nutr. 2016 Dec;104(6):1534-1544. doi: 10.3945/ajcn.116.137919. Epub 2016 Oct 26. PMID 27797709